CLINICAL TRIAL: NCT05893459
Title: Beneficial or Fostering Future Struggles (B.F.F.s)? Characterizing the Role of Friends in Adolescent Development
Brief Title: Beneficial or Fostering Future Struggles (B.F.F.s)? Characterizing the Role of Friends in the Development of 13- to 17-Year-Old Adolescents
Acronym: BFFs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michelle P. Brown, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00125559; R00HD103958 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-06-08 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Child Maltreatment; Interpersonal Relations; Victimisation; Psychopathology; Electrocardiography
Keywords: Adolescents; Teenagers; Teens; Youth; Friendship; Friends; Mental Health; Psychopathology; Psychological Trauma; Childhood Trauma; Child Abuse; Child Neglect; Child Maltreatment; Psychophysiology; Respiratory Sinus Arrhythmia; Longitudinal Studies
MeSH Terms: conditions — Psychological Well-Being; Psychological Trauma; Arrhythmia, Sinus

STUDY DESIGN:
Intervention Model Description: Debrief - Following exposure to a laboratory stressor, adolescent participants will be randomly assigned to either debrief their experience with a friend or sit by themselves (standard procedure) while their psychophysiological reactivity is recorded using an electrocardiogram (ECG).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debrief (Experimental): Following exposure to a laboratory stressor, participants in this arm will debrief their experience with a friend for 5 minutes while their psychophysiological reactivity is recorded using an electrocardiogram (ECG). Their interaction will be audio and video recorded for later observational coding of their friend's validating and invalidating behaviors during the conversation.
  Interventions: Behavioral: Debrief
- No Debrief (No Intervention): Following exposure to a laboratory stressor, participants in this arm will sit by themselves while their psychophysiological reactivity is recorded using an electrocardiogram (ECG).

INTERVENTIONS:
Behavioral: Debrief — Post-Stressor Discussion with a Friend
  Arms: Debrief

SUMMARY:
The goal of this clinical trial is to investigate how the friendship experiences of maltreated (i.e., abused and/or neglected) and non-maltreated adolescents differentially influence their risk for adverse outcomes. The main questions it aims to answer are:

1. How do the friendships of maltreated adolescents differ from those of non-maltreated adolescents?
2. Which friendship experiences influence the associations between maltreatment and ability to regulate stress, as well as future mental health difficulties and revictimization?

Participants will:

* Attend the initial study visit on the campus of the University of South Carolina with their primary caregiver and a best friend during which they will:

  * Complete study questionnaires
  * Be connected to a device that records their physical ability to manage stress
  * Complete a task during which they will be audio and video recorded and complete a brief assessment rating how they are feeling at different times during task completion
  * Depending on which research group they are placed in, be assigned to discuss their experience doing this task with their friend (intervention group) or sit quietly in a room for 5 minutes (comparison group)
* The follow-up study visit will involve completion of study questionnaires online or via mail 6 months later

Additionally, the participant's caregiver and friend will complete study questionnaires.

Researchers will compare the intervention group (debriefs with a friend) and comparison group (sits quietly for 5 minutes) to see if the presence of and discussion with the friend influences their physical ability to regulate stress and future outcomes.

DETAILED DESCRIPTION:
When potential participants indicate interest in the study, participants and caregivers will first complete pre-screening measures to inquire about child welfare system involvement and determine eligibility. If eligible, they will be contacted for scheduling and the caregiver will be administered a brief trauma screen to determine maltreatment status and adolescents will identify a friend to accompany them to the assessment. The study team will then schedule a laboratory visit and participants will be instructed to bring their friend and caregiver. The participant, caregiver, friend, and friend's caregiver will then complete consent and assent procedures. The adolescent and friend will then complete measures related to their friendship experiences as applicable prior to administration of a laboratory stressor, the Trier Social Stress Test (TSST). Adolescents will then be randomly assigned to discuss their TSST experience with their friend or wait in a room by themselves (standard TSST procedure) using a blocked randomization procedure to balance the two groups on maltreatment status and gender, thereby reducing bias and confounding that may be attributable to these factors. This randomization will be performed using a computer algorithm with randomly selected block sizes of 4, 6, and 8. There will be twice as many participants being randomized to debrief with a friend as are randomized to the standard TSST procedure. This is done for several reasons. First, this is done to maximize power for examining the potential moderating effect of friendship experiences (i.e., validating and invalidating responses from friends following adolescents' stressor exposure) that can only be assessed if participants are randomized to this condition. Second, the standard procedure has already been extensively implemented and studied in developmental/clinical research, including with children who have experienced maltreatment and other forms of adversity along with children's/adolescent's psychophysiological reactivity in response to undergoing this stressor. Thus, it is important to collect more novel data regarding how the presence of a friend and their accompanying responses toward the participant influence adolescents' ability to recover following this stressor.

Their psychophysiological, or or respiratory sinus arrhythmia (RSA) activity, will be measured using an electrocardiogram (ECG) before, during, and after the TSST during either the 5-minute post-TSST discussion with their friend or a 5-minute period during which the adolescent is by themselves. For those assigned to debrief with a friend, validating and invalidating responses of the friend toward the adolescent participant will be observed and coded. Participants will be followed up six months later at Time 2 (T2) and adolescents and their parents will complete additional measures related to friendship, psychopathology, and revictimization experiences, online or via mail, if needed.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 17 years old at first study visit
* Qualify as either maltreated (endorses history of maltreatment - physical abuse, sexual abuse, emotional maltreatment, or neglect and/or has substantiated record of child maltreatment per Department of Social Services [DSS] records) or non-maltreated (denies history of maltreatment and/or no substantiated record of child maltreatment per DSS records)
* Parent participating in the study visit is a non-offending caregiver (no record of substantiated maltreatment against the adolescent participant)
* Participant identifies a best friend who is not a sibling or previous/current romantic partner who can accompany them to the study visit
* Participant, caregiver, and friend are fluent in written and spoken English

Exclusion Criteria:

* <13 or >17 at time of first study visit
* No available non-offending parent or guardian/caregiver to participate in the study
* No best friend identified to accompany the participant to the study
* Participant, caregiver, or friend is not fluent in written and spoken English

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory sinus Arrhythmia (RSA) activity | Baseline
  RSA activity, including resting RSA (prior to Trier Social Stress Test [TSST] procedure), RSA reactivity (difference between RSA activity during stressor exposure and resting RSA), and RSA recovery (difference between RSA activity during 5 minutes post stressor exposure whether during debriefing with friend or in isolation and RSA activity during stressor exposure).
Youth Self Report (YSR) | 6 Month Follow Up from Baseline
  YSR, which is completed by the adolescent and assesses the participant's internalizing (e.g., anxious, depressed) and externalizing (e.g., aggression, rule-breaking behavior) symptoms. Scale scores are reported for Internalizing and Externalizing symptoms and higher scores indicate greater symptoms and a worse outcome. Possible raw scores range from 0 to 62 for Internalizing Symptoms and 0 to 60 for Externalizing Symptoms. Raw scores are transformed to standardized T scores normed by age and gender ranging from 26 to 100 for Internalizing and 25 to 100 for Externalizing.
Child Behavior Checklist (CBCL) | 6 Month Follow-Up from Baseline
  CBCL, which is a parallel form to the YSR completed by the caregiver and assesses the participant's internalizing (e.g., anxious, depressed) and externalizing (e.g., aggression, rule-breaking behavior) symptoms. Scale scores are reported for Internalizing and Externalizing symptoms and higher scores indicate greater symptoms and a worse outcome. Possible raw scores range from 0 to 62 for Internalizing Symptoms and 0 to 66 for Externalizing Symptoms. Raw scores are transformed to standardized T scores normed by age and gender ranging from 31 to 100 for Internalizing and 30 to 100 for Externalizing.
University of California, Los Angeles Posttraumatic Stress Disorder Reaction Index (UCLA PTSD-RI) for the Diagnostic and Statistical Manual of Mental Disorders -5th Edition (DSM-5) Total Score | 6 Month Follow-Up from Baseline
  UCLA PTSD Reaction Index for the DSM-5, which is completed by the adolescent participant and their caregiver and provides an overall PTSD symptom based on DSM-5 criteria. Total score ranges from 0 to 80 and higher scores indicating greater symptoms and a worse outcome.
Juvenile Victimization Questionnaire (JVQ) total score | 6 Month Follow-Up from Baseline
  JVQ, which is completed by the adolescent participant and assesses experiences with five areas of youth victimization (i.e., conventional crime, peer and sibling victimization, maltreated, sexual victimization, and witnessing and indirect victimization) that has occurred within the past six months since the first study visit. A count of total experiences endorsed ranging from 0 to 34 is computed with a higher score indicating more victimization and a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request by the PI, in a format that protects the privacy and anonymity of study participants. Specifically, even though the final dataset will be stripped of identifiers prior to release for sharing, we believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will be shared via a secure institutionally supported data archive (e.g., Microsoft One Drive and/or Box).
Time Frame: Starting 6 months after publication
Access Criteria: Data will be made available upon request by the PI, in a format that protects the privacy and anonymity of study participants. We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will be shared via a secure institutionally supported data archive (e.g., Microsoft One Drive and/or Box). PI will review all data sharing requests.

REFERENCES:
- [Background] Parker, J. G., Rubin, K. H., Erath, S. A., Wojslawowicz, J. C., & Buskirk, A. A. (2006). Peer relationships, child development, and adjustment: A developmental psychopathology perspective. In D. Cicchetti & D. J. Cohen (Eds.), Developmental psychopathology: Theory and method (pp. 419-493). John Wiley & Sons Inc; US.
- [Background] Mueller, E., & Silverman, N. (1989). Peer relations in maltreated children. In D. Cicchetti & Carlson, Vicki (Eds.), Child maltreatment: Theory and research on the causes and consequences of child abuse and neglect. (pp. 529-578). https://doi.org/10.1017/CBO9780511665707.018
- [Background] Prinstein, M. J., & Giletta, M. (2016). Peer relations and developmental psychopathology. In D. Cicchetti (Ed.), Developmental psychopathology: Theory and method (pp. 527-579). John Wiley & Sons Inc; US.
- [Background] Hartup, W. W., & Stevens, N. (1997). Friendships and adaptation in the life course. Psychological Bulletin, 121(3), 355-370. https://doi.org/10.1037/0033-2909.121.3.355
- [Background] Calhoun CD, Helms SW, Heilbron N, Rudolph KD, Hastings PD, Prinstein MJ. Relational victimization, friendship, and adolescents' hypothalamic-pituitary-adrenal axis responses to an in vivo social stressor. Dev Psychopathol. 2014 Aug;26(3):605-18. doi: 10.1017/S0954579414000261. PMID 25047287
- [Background] Doom JR, Doyle CM, Gunnar MR. Social stress buffering by friends in childhood and adolescence: Effects on HPA and oxytocin activity. Soc Neurosci. 2017 Feb;12(1):8-21. doi: 10.1080/17470919.2016.1149095. Epub 2016 Feb 25. PMID 26899419
- [Background] Hodges EV, Boivin M, Vitaro F, Bukowski WM. The power of friendship: protection against an escalating cycle of peer victimization. Dev Psychol. 1999 Jan;35(1):94-101. doi: 10.1037//0012-1649.35.1.94. PMID 9923467
- [Background] Desir MP, Karatekin C. Characteristics of Disclosing Childhood Victimization and Risk of Revictimization in Young Adulthood. J Interpers Violence. 2021 Nov;36(21-22):NP12225-NP12251. doi: 10.1177/0886260519889932. Epub 2019 Dec 3. PMID 34755561
- [Background] Allen EK, Desir MP, Shenk CE. Child maltreatment and adolescent externalizing behavior: Examining the indirect and cross-lagged pathways of prosocial peer activities. Child Abuse Negl. 2021 Jan;111:104796. doi: 10.1016/j.chiabu.2020.104796. Epub 2020 Nov 12. PMID 33189371
- [Background] Brown, M. P. (2019). Developmental Pathways from Childhood Maltreatment to Adolescent Psychopathology, Substance Use, and Revictimization. http://conservancy.umn.edu/handle/11299/206323
- [Background] Merritt DH, Snyder SM. Correlates of optimal behavior among child welfare-involved children: Perceived school peer connectedness, activity participation, social skills, and peer affiliation. Am J Orthopsychiatry. 2015 Sep;85(5):483-94. doi: 10.1037/ort0000091. PMID 26460707
- [Background] Ezzell CE, Swenson CC, Brondino MJ. The relationship of social support to physically abused children's adjustment. Child Abuse Negl. 2000 May;24(5):641-51. doi: 10.1016/s0145-2134(00)00123-x. PMID 10819096
- [Background] Folger, S. F., & Wright, M. O. (2013). Altering risk following child maltreatment: Family and friend support as protective factors. Journal of Family Violence, 28(4), 325-337. https://doi.org/10.1007/s10896-013-9510-4
- [Background] Powers A, Ressler KJ, Bradley RG. The protective role of friendship on the effects of childhood abuse and depression. Depress Anxiety. 2009;26(1):46-53. doi: 10.1002/da.20534. PMID 18972449
- [Background] Long SJ, Evans RE, Fletcher A, Hewitt G, Murphy S, Young H, Moore GF. Comparison of substance use, subjective well-being and interpersonal relationships among young people in foster care and private households: a cross sectional analysis of the School Health Research Network survey in Wales. BMJ Open. 2017 Feb 20;7(2):e014198. doi: 10.1136/bmjopen-2016-014198. PMID 28219960
- [Background] Segura A, Pereda N, Guilera G, Hamby S. Resilience and psychopathology among victimized youth in residential care. Child Abuse Negl. 2017 Oct;72:301-311. doi: 10.1016/j.chiabu.2017.08.019. Epub 2017 Sep 1. PMID 28866317
- [Background] U.S. Department of Health and Human Services, Administration for Children and Families, Administration on Children, Youth and Families, Children's Bureau. (2019). Child Maltreatment 2017. Retrieved from https://www.acf.hhs.gov/cb/research-data-technology/ statistics-research/child-maltreatment
- [Background] Cicchetti, D., & Toth, S. L. (2016). Child maltreatment and developmental psychopathology: A multilevel perspective. In D. Cicchetti (Ed.), Developmental psychopathology: Vol. Maladaptation and Psychopathology (pp. 1-55). https://doi.org/10.1002/9781119125556.devpsy311
- [Background] Wang, C.-T., & Holton, J. (2007). Total estimated cost of child abuse and neglect in the United States. Prevent Child Abuse America Chicago, IL.
- [Background] Parker, J. G., & Herrera, C. (1996). Interpersonal processes in friendship: A comparison of abused and nonabused children's experiences. Developmental Psychology, 32(6), 1025-1038. http://dx.doi.org/10.1037/0012-1649.32.6.1025
- [Background] Cicchetti D. Annual Research Review: Resilient functioning in maltreated children--past, present, and future perspectives. J Child Psychol Psychiatry. 2013 Apr;54(4):402-22. doi: 10.1111/j.1469-7610.2012.02608.x. Epub 2012 Aug 28. PMID 22928717
- [Background] Cicchetti D, Rogosch FA. The role of self-organization in the promotion of resilience in maltreated children. Dev Psychopathol. 1997 Fall;9(4):797-815. doi: 10.1017/s0954579497001442. PMID 9449006
- [Background] Desir, M. P. & Karatekin, C. (2020). Interpersonal factors influencing risk for revictimization in two samples of young adults. Journal of Child Custody, 17(2), 89-115. https://doi.org/10.1080/26904586.2020.1751015
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Roussos A, Goenjian AK, Steinberg AM, Sotiropoulou C, Kakaki M, Kabakos C, Karagianni S, Manouras V. Posttraumatic stress and depressive reactions among children and adolescents after the 1999 earthquake in Ano Liosia, Greece. Am J Psychiatry. 2005 Mar;162(3):530-7. doi: 10.1176/appi.ajp.162.3.530. PMID 15741470
- [Background] Barnett, D., Manly, J. T., & Cicchetti, D. (1993). Defining child maltreatment: The interface between policy and research. In D. Cicchetti & S. L. Toth (Eds.), Child abuse, child development, and social policy. Ablex
- [Background] Shenk, C. E., & Fruzzetti, A. E. (2011). The impact of validating and invalidating responses on emotional reactivity. Journal of Social and Clinical Psychology; New York, 30(2), 163-183. http://dx.doi.org/10.1521/jscp.2011.30.2.163
- [Background] Shenk, C. E., & Fruzzetti, A. E. (2014). Parental validating and invalidating responses and adolescent psychological functioning: An observational study. The Family Journal, 22(1), 43-48. https://doi.org/10.1177/1066480713490900
- [Background] Furman, W., & Buhrmester, D. (1985). Children's perceptions of the personal relationships in their social networks. Developmental Psychology, 21(6), 1016-1024. http://dx.doi.org/10.1037/0012-1649.21.6.1016
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Achenbach, T. M. (1991). Integrative guide for the 1991 CBCL/4-18, YSR, and TRF Profiles. Department of Psychiatry, University of Vermont.
- [Background] Davidian, M., & Giltinan, D. M. (1995). Nonlinear models for repeated measurement data (Vol. 62). Chapman & Hall.
- [Background] Briere J, Johnson K, Bissada A, Damon L, Crouch J, Gil E, Hanson R, Ernst V. The Trauma Symptom Checklist for Young Children (TSCYC): reliability and association with abuse exposure in a multi-site study. Child Abuse Negl. 2001 Aug;25(8):1001-14. doi: 10.1016/s0145-2134(01)00253-8. PMID 11601594
- [Background] Finkelhor D, Hamby SL, Ormrod R, Turner H. The Juvenile Victimization Questionnaire: reliability, validity, and national norms. Child Abuse Negl. 2005 Apr;29(4):383-412. doi: 10.1016/j.chiabu.2004.11.001. PMID 15917079
- [Background] Brown MP, Ng R, Lisle J, Koenig M, Sannes D, Rogosch F, Cicchetti D. Mind-mindedness in a high-risk sample: Differential benefits for developmental outcomes based on child maltreatment. Dev Psychol. 2023 Jun;59(6):1126-1135. doi: 10.1037/dev0001506. Epub 2023 Jan 5. PMID 36603122